CLINICAL TRIAL: NCT01482052
Title: A Double-Blind, Randomized, Controlled, Two Arm Phase 1 Clinical Trial of the Safety and Immunogenicity of Group A, C, Y & W-135 Meningococcal Polysaccharide DT Conjugate Vaccine: NmVac4-A/C/Y/W-135-DT™
Brief Title: Safety Study of Group A, C, Y & W-135 Meningococcal Polysaccharide Diphtheria Toxoid Conjugate Vaccine for Meningitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: JN-International Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JN-NM-001
Record Dates: First submitted 2011-11-23; First posted 2011-11-30 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Meningococcal Meningitis; Meningococcal Infections
Keywords: Central Nervous System Infections; Meningitis; toxoid; Meningococcal vaccine; conjugate vaccines
MeSH Terms: conditions — Meningitis, Meningococcal; Meningococcal Infections; Central Nervous System Infections; Meningitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test Vaccine (Experimental): NmVac4-A/C/Y/W-135-DT™ conjugate vaccine
  Interventions: Biological: meningococcal meningitis conjugate vaccine, quadrivalent
- US Licensed Vaccine (Active Comparator): Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine
  Interventions: Biological: meningococcal meningitis conjugate vaccine, quadrivalent

INTERVENTIONS:
Biological: meningococcal meningitis conjugate vaccine, quadrivalent — NmVac4-A/C/Y/W-135-DT™conjugate is a vaccine in liquid form composed of purified polysaccharides (PS) conjugated to diphtheria toxoid. Single intramuscular 0.5 mL dose contains 4 µg each Serogroup A, C, W-135, Y PS conjugated to approximately 16 µg total diphtheria toxoid.
  Other Names: NmVac4-A/C/Y/W-135-DT™
  Arms: Test Vaccine
Biological: meningococcal meningitis conjugate vaccine, quadrivalent — Meningococcal (Groups A,C,Y and W-135-DT) Polysaccharide Conjugate Vaccine 0.5 mL dose, intramuscular. Single dose contains 4 µg each Serogroup A, C, W-135, Y PS conjugated to approximately 48 µg total diphtheria toxoid.
  Arms: US Licensed Vaccine

SUMMARY:
The purpose of this study is to evaluate the safety of a new conjugate vaccine, NmVac4-A/C/Y/W-135-DT, compared to the safety of a similar, licensed meningococcal A/C/Y/W-135-DT conjugate vaccine. The investigators will also evaluate the production of antibodies to of NmVac4-A/C/Y/W-135-DT™ conjugate vaccine compared to the licensed vaccine, as a measure of vaccine effectiveness.

DETAILED DESCRIPTION:
Meningococcal disease is a potentially life-threatening bacterial infection. The disease most commonly is expressed as either meningococcal meningitis, an inflammation of the membranes surrounding the brain and spinal cord, or meningococcemia, the presence of bacteria in the blood. The most common symptoms include high fever, headache, neck stiffness, confusion, nausea, vomiting, lethargy, and rash. If not treated the disease can progress rapidly and can lead to shock and death, often within hours of the onset of symptoms. Neisseria meningitidis capsular polysaccharides are poor immunogens. However, conjugation of bacterial polysaccharides to immunogenic carrier proteins generally results in conjugates that induce strong anti-polysaccharide T-helper cell dependent immune responses, creating a longer-lasting immune response and thus protection against meningococcal infection. This study compares safety and antibody production induced by one intramuscular injection of either NmVac4-A/C/Y/W-135-DT or a licensed meningococcal A/C/Y/W-135-DT conjugate vaccine. Participants will attend a screening visit up to 4 weeks prior to Day 0, then will attend study visits for 8 weeks. There will be a study phone call at Days 2-3, then a post-study telephone call to subjects to assess safety at 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent and comply with all aspects of the evaluation after the nature of the study is explain
* For the purpose of this study, a healthy volunteer is defined as healthy male or female, with no significant chronic conditions
* Age 18 to 50 years old
* Either gender. Abstinence or use of contraception during the eight weeks after vaccination will be required for non menopausal (< two years post-menopause) or non surgically sterile women
* Persons with antibody titer(s) of <2 µg/mL to serogroup(s) A, C, Y, or W-135 polysaccharides as measured by ELISA

Exclusion Criteria:

* Age less than 18 years or over 50 years.
* History of Guillain-Barré syndrome (GBS).
* Pregnancy or lactation.
* History of meningococcal meningitis.
* History of invasive (clinical or laboratory diagnosis) meningococcal disease.
* History of meningococcal meningitis vaccination.
* Screening laboratory abnormalities (in the opinion of the Investigator) that would raise safety concerns for participation in the study.
* Use of immunosuppressive drugs within 30 days prior to study enrollment, not including topical or inhaled steroids/cytotoxic agents.
* History of anaphylactic shock, asthma, urticaria, or other allergic or hypersensitivity reactions following vaccination.
* History of severe allergic disorders or autoimmune connective tissue disorders, including rheumatoid arthritis. A high sensitivity C-Reactive Protein (CRP) test at screening will be used as part of the assessment of autoimmune disorders by the Principal Investigator.
* Use of systemic antibiotics within 72 hours prior to study enrollment.
* History of cirrhosis.
* Positive results of testing for HepBsAg, Hepatitis C or HIV-1 or HIV-2 antibodies.
* Positive results of drug screen (amphetamine, THC, cocaine).
* Persons with antibody titer(s) of >2 µg/mL to serogroup (s) A, C, Y, or W 135 as measured by ELISA.
* Unable to understand all of the study requirements.
* Prisoners.
* Participation in a clinical trial in the last three months.
* History of any serious chronic medical or psychiatric illnesses.
* History of significant head trauma, alcohol or substance abuse or other medical illnesses that could cause a neurological deficit (e.g., cerebro-vascular disease) .
* Chronic medication use that, in the opinion of the Investigator, may influence or bias the clinical outcome of the trial.
* Individuals will be excluded from participation in this trial if they are judged by the Principal Investigator as having a significant impairment in their capacity for judgment or reasoning that compromise their ability to make decisions in their best interest.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Adverse Reactions | up to 6 months
  local and systemic rates throughout the course of the study

SECONDARY OUTCOMES:
Immune Response | 4 and 8 weeks after injection
  Antibody titers

CONTACTS AND LOCATIONS:
Overall Officials: Sudesh Nagavalli, MD, Principal Investigator
Locations (1):
- Kings Cardiology Group, Hanford, California, United States